CLINICAL TRIAL: NCT03019809
Title: A Trial of Plerixafor With G-CSF as Additional Agents in Conditioning Regimen for Prevention of Graft Failure After Transplantation With TCR Alpha/Beta Grafts Depletion in Patients With Wiskott-Aldrich Syndrome.
Brief Title: A Trial of Plerixafor/G-CSF as Additional Agents for Conditioning Before TCR Alpha/Beta Depleted HSCT in WAS Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WAS_PG 2016
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Wiskott-Aldrich Syndrome; Hematopoietic Stem Cell Transplantation; Graft Failure
MeSH Terms: conditions — Wiskott-Aldrich Syndrome | interventions — Granulocyte Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Plerixafor/G-CSF for HSCT conditioning (Experimental): Myeloablative conditioning regimen with Plerixafor and G-CSF as addition agents before stem cell transplantation in WAS patients.
  Interventions: Biological: G-CSF for Conditioning before HSCT.; Biological: Plerixafor for Conditioning before HSCT.

INTERVENTIONS:
Biological: G-CSF for Conditioning before HSCT. — Mobilization of hematopoietic stem (HSC) into circulation
Biological: Plerixafor for Conditioning before HSCT. — Directed inhibition of CXC chemokine receptor type 4 (CXCR4) for opening enough BM niches for adequate donor HSC engraftment.

SUMMARY:
Treatment Study to assess of safety and efficiency of conditioning with Plerixafor and G-CSF as additional agents for prevention of graft failure after transplantation with TCR alpha/beta grafts depletion in patient with Wiskott-Aldrich syndrome.

DETAILED DESCRIPTION:
Severe graft dysfunction, such as the degree of donor chimerism predominantly in the myeloid compartment is one of major problem in patients with Wiskott-Aldrich syndrome (WAS), especially after hematopoietic stem cell transplantation (HSCT) from alternative donor. It often leads to the development of severe thrombocytopenia or even transplants rejection. In this study the hypothesis is that the use of plerixafor and G-CSF as additional agents in conditioning regimen would offers advantages due to lowing risk of mixed chimerism after HSCT. This effect is based on the fact that simultaneous use of plerixafor with G-CSF is efficient in inducing stem cell release and opening of bone marrow (BM) niches. Moreover, stem cell release probably leads to liberation of host stem cells from the anti-apoptotic effects of the BM stroma for the more powerful effect of chemotherapy.

In this study, the investigators use TCR alpha/beta grafts depletion of the grafts as basic technology for HSCT from haploidentical and unrelated donors approved in Institution.

Thus, the purpose of this study is to evaluate the safety and efficiency of myeloablative conditioning with Plerixafor and G-CSF as additional agents for prevention of graft failure after transplantation with TCR alpha/beta grafts depletion in patients with Wiskott-Aldrich syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 1 months and < 19 years
* Patients diagnosed with Wiskott-Aldrich syndrome eligible for an allogeneic transplantation and lacking a related HLA-matched donor
* Lansky/Karnofsky score > 40, WHO > 4
* Signed written informed consent

Exclusion Criteria:

* Dysfunction of liver (ALT/AST > 5 times normal value, or bilirubin > 3 times normal value), or of renal function (creatinine clearance < 30 ml / min)
* Severe cardiovascular disease (arrhythmias requiring chronic treatment, congestive heart failure or left ventricular ejection fraction <40%)
* Serious concurrent uncontrolled medical disorder
* Lack of parents' informed consent.

Ages: 1 Month to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Event free survival (EFS) | 24 months
  The EFS probability compared with historical control. We mean event as patient's death, second transplantation or persistence of severe thrombocytopenia

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
  The OS probability compared with historical control.
Percentage of patients with full/mixed donor chimerism | 12 months
  Evaluation of the percentage of patients with the full/mixed donor chimerism (whole blood and CD3+ lineage). In addition, patients will be divided in accordance with % of donors cells: >95%; 50%-95%; 10%-49%; <10%. All data will be compared with historical control
Transplant related mortality (TRM) | 24 months
  The TRM probability compared with historical control.
Severe thrombocytopenia (ST) | 24 months
  The ST probability after HSCT compared with historical control
Autoimmune complications (AC) | 24 months
  The AC probability after HSCT compared with historical control
Acute Graft Versus Host Diseases (aGVHD) | 12 months
  Cumulative Incidence and severity of aGVHD
Chronic Graft Versus Host Diseases (cGVHD) | 24 months
  Cumulative Incidence and severity of cGVHD
Plerixafor related complications (PRC) | 2 week
  PRC: severity, features, incidence

CONTACTS AND LOCATIONS:
Overall Officials: Alexei Maschan, Professor, Study Chair — Dmitry Rogachev Federal Research and Clinical Centre of Paediatric Haematology, Oncology and Immunology; Dmitry Balashov, Principal Investigator — Dmitry Rogachev Federal Research and Clinical Centre of Paediatric Haematology, Oncology and Immunology
Locations (1):
- Dmitry Rogachev Federal Research and Clinical Centre of Paediatric Haematology, Oncology and Immunology, Moscow, Russia

REFERENCES:
- [Derived] Balashov D, Laberko A, Shcherbina A, Trakhtman P, Abramov D, Gutovskaya E, Kozlovskaya S, Shelikhova L, Novichkova G, Maschan M, Rumiantsev A, Maschan A. A Conditioning Regimen with Plerixafor Is Safe and Improves the Outcome of TCRalphabeta+ and CD19+ Cell-Depleted Stem Cell Transplantation in Patients with Wiskott-Aldrich Syndrome. Biol Blood Marrow Transplant. 2018 Jul;24(7):1432-1440. doi: 10.1016/j.bbmt.2018.03.006. Epub 2018 Mar 14. PMID 29550630